CLINICAL TRIAL: NCT00468000
Title: Use of Ixmyelocel-T (Formerly TRC Autologous Bone Marrow Cells) in Patients With Peripheral Arterial Disease to Treat Critical Limb Ischemia
Brief Title: Use of Ixmyelocel-T (Formerly Vascular Repair Cells [VRC]) in Patients With Peripheral Arterial Disease to Treat Critical Limb Ischemia
Acronym: RESTORE-CLI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABI-55-0610-1
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Critical Limb Ischemia; Ischemia; Peripheral Vascular Disease; ixmyelocel-T
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Ischemia; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ixmyelocel-T (Experimental): The treatment arm of the study will receive injections of the study cellular product.
  Interventions: Biological: Ixmyelocel-T
- Placebo (Placebo Comparator): The control arm of the study will receive placebo injections.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ixmyelocel-T — IM injection
  Arms: Ixmyelocel-T
Biological: Placebo — IM Injection
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and efficacy of autologous Vascular Repair Cells (VRC) for patients with peripheral arterial disease as a treatment for critical limb ischemia.

The double-blind study is expected to enroll 150 patients, randomized into two patient groups. The treatment group will receive intramuscular (IM) injections of the VRCs into the affected limb; the control group will receive intramuscular injections with an electrolyte solution (without cells). Both groups will receive the standard of care appropriate for their medical condition.

DETAILED DESCRIPTION:
The study will assess the safety and ability of Aastrom TRC autologous bone marrow cells to restore peripheral blood flow affected by critical limb ischemia.

Peripheral arterial disease (PAD), also known as Peripheral Vascular Disease (PVD), occurs when peripheral arteries are damaged by arterial hypertension and/or by the formation of atherosclerotic plaques. PAD is a chronic disease that progressively constricts arterial circulation of limbs. The term critical limb ischemia (CLI) is used for all patients with chronic ischemia rest pain, ulcers, or gangrene in limbs attributable to objectively proven PAD. These sequelae represent the end stage of PAD. PAD is associated with several other clinical conditions, i.e. hypertension, cardiovascular disease, hyperlipidemia, diabetes, tobacco use, obesity and stroke.

The double-blind study is expected to enroll 150 patients, randomized into two patient groups. The treatment group will receive intramuscular injections of the TRC product into the affected limb; the control group will receive intramuscular injections with an electrolyte solution (without cells). Both groups will receive the standard of care appropriate for their medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-90 years of age
* Diagnosis of CLI
* Infrainguinal occlusive disease, without options for revascularization
* No surgical interventions planned
* Life expectancy of 2 years
* Normal organ and marrow function
* Patients with controlled blood pressure (≤ 180/110 mmHg) and established anti-hypertensive therapy
* Established anti-platelet therapy

Exclusion Criteria:

* Poorly controlled diabetes mellitus (hemoglobin A1c [HbA1c] > 10%)
* Aortoiliac disease with > 50% stenosis
* Wounds with severity greater than Grade 3 on the Wagner Scale
* Any known failed ipsilateral revascularization within 2 weeks of enrollment
* Previous amputation of the talus, or above in the target limb
* Life-threatening ventricular arrhythmia; unstable angina; or, myocardial infarction within 4 weeks of enrollment
* Severe congestive heart failure (CHF) (i.e. New York Heart Association [NYHA] Stage IV)
* Receiving treatment with hematopoietic growth factors
* Infection of the involved extremity(ies)
* Active wet gangrenous tissue
* Require uninterruptible anticoagulation therapy
* Blood clotting disorder
* Cancer
* End stage renal disease requiring dialysis for more than 6 months prior to enrollment
* Pregnant or lactating
* Having received medication for thrombolytic therapy (e.g. rTPA or other enzymatic clot busters) within 30 days prior to enrollment
* Undergoing hyperbaric oxygen treatment within 2 weeks of enrollment
* Concomitant wound treatments with growth factors or tissue engineered products
* Receiving anti-angiogenic drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety of TRCs in patients with CLI(key safety parameters include vital signs, physical exams, laboratory results, assessment of aspiration and injection sites, adverse events, major amputations, wounds presence(size and grading using the Wagner scale) | throughout trial

SECONDARY OUTCOMES:
Composite efficacy endpoint assessing time to treatment failure(failure defined as major amputation, doubling of wound size, and new gangrene) | Day 7 and Months 3, 6, 9, 12
Percentage of patients failing treatment | Day 7, and Months 3,6,9, and 12
Time to major amputation | Day 7 and Month 3, 6, 9, and 12
Percentage of patients undergoing major amputation | Day 7 and Months 3, 6, 9, 12
Incidence of revascularization interventions throughout duration of study | Day 7 and Months 3,6,9,12
Incidence of bypass surgery for patients throughout duration of study | Day 7 and Months 3,6,9,12
Healing of all wounds in the target limb | Day 7 and Months 3,6,9,12
Ankle and/or toe pressure and ankle brachial pressure index and/or toe brachial index | Day 7 and Months 3,6,9,12
Pain, as measured by visual analog scale(VAS) | Day 7 and Months 3,6,9,12
The King's College Vascular Quality of Life Questionnaire | Baseline and Months 6 and 12
Walking distance as measured by six-minute walk test(with or without walking device) | Baseline and Month 12
Concurrent Meds for trends | Day 7 and Months 3, 6, 9, 12

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Comerota, MD, Principal Investigator — Jobst Vascular Center
Locations (20):
- United States (20):
  - Cardiology, P.C., Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - Malcolm Randall Veterans Administration Medical Center, part of the North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - University of Miami/Miller School of Medicine, Miami, Florida
  - Loyola University Stritch School of Medicine, Maywood, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - The Care Group, LLC, Indianapolis, Indiana
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Vascular Research Center, Flint, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Memorial Center, Lebanon, New Hampshire
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Jobst Vascular Center, Toledo, Ohio
  - Oklahoma University, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Peripheral Vascular Associates, San Antonio, Texas
  - Scott and White Hospital, Temple, Texas

REFERENCES:
- [Result] Powell RJ, Marston WA, Berceli SA, Guzman R, Henry TD, Longcore AT, Stern TP, Watling S, Bartel RL. Cellular therapy with Ixmyelocel-T to treat critical limb ischemia: the randomized, double-blind, placebo-controlled RESTORE-CLI trial. Mol Ther. 2012 Jun;20(6):1280-6. doi: 10.1038/mt.2012.52. Epub 2012 Mar 27. PMID 22453769
- [Result] Powell RJ, Comerota AJ, Berceli SA, Guzman R, Henry TD, Tzeng E, Velazquez O, Marston WA, Bartel RL, Longcore A, Stern T, Watling S. Interim analysis results from the RESTORE-CLI, a randomized, double-blind multicenter phase II trial comparing expanded autologous bone marrow-derived tissue repair cells and placebo in patients with critical limb ischemia. J Vasc Surg. 2011 Oct;54(4):1032-41. doi: 10.1016/j.jvs.2011.04.006. Epub 2011 Jul 31. PMID 21684715
- [Derived] Moazzami B, Mohammadpour Z, Zabala ZE, Farokhi E, Roohi A, Dolmatova E, Moazzami K. Local intramuscular transplantation of autologous bone marrow mononuclear cells for critical lower limb ischaemia. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD008347. doi: 10.1002/14651858.CD008347.pub4. PMID 35802393